CLINICAL TRIAL: NCT06262828
Title: Harnessing Evidence And Real-world Data To Improve Cardiovascular Health and Services (HEARTWISE) - The Personalised - CARdiovascular DIsease Risk Assessment for Chinese (P-CARDIAC) Real World Evidence Study - Population-based Study
Brief Title: HEARTWISE - P-CARDIAC for Chinese: Population-based Study
Acronym: HEARTWISE
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Sze Ling Celine Chui, Assistant Professor, The University of Hong Kong
Other Study IDs: CIRB-2024-240-3
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; CVD
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease (CVD) is one of the prominent diseases that affect many people. One cost-effective solution is to identify people at higher risk of CVD by CVD risk prediction model. China-PAR, TRS-2P, and SMART2 are common risk prediction models for prevention. However, these risk scores were mostly based on the routinely self-check health information and multivariable regression without time-varying consideration. Investigators developed a Machine Learning (ML) based risk prediction model, Personalized CARdiovascular DIsease risk Assessment for Chinese (P-CARDIAC) among a predominantly Chinese population in Hong Kong to estimates the 10 years of secondary recurrent CVD risk for the high-risk individuals. The study objective is to evaluate the accuracy of the P-CARDIAC performance in practice among a large-scale Hong Kong population in medicine specialist outpatient clinic (SOPC) and cardiac clinic. The results will reassure cardiologists that the P-CARDIAC risk score is sensitive to the heart disease symptoms. Investigators anticipate that the results may help to facilitate P-CARDIAC in clinical setting and provide more practical information with the development of P-CARDIAC.

DETAILED DESCRIPTION:
This study has two parts to conduct for different outcomes.

Part one is a prospective population-based cohort study. Investigators hypothesize that patients with a higher frequency or larger number of types of cardiac event symptoms are likely to have a higher P-CARDIAC risk score. The correlation between P-CARDIAC risk score and the increasing in number of types and in number of times a patient reported to have heart disease symptoms, e.g. chest pain, shortness of breath, fatigue, swelling in legs, ankles or feet will be examined. The results reassure cardiologists that the P-CARDIAC risk score is sensitive to the heart disease symptoms. Patients who are at a higher risk of recurrent CVD event are likely to have more medications and to have a sooner follow up appointment. At such, investigators also hypothesize a positive relationship between P-CARDIAC risk score and the number of class of medications prescribed and a negative correlation between P-CARDIAC risk score and the time to next SOPC follow up appointment.

Part two of the study will involve Delphi technique to determine P-CARDIAC risk thresholds with reference to current clinical management guideline such as American Heart Association (AHA)/American College of Cardiology (ACC) Multisociety Guideline (AHA/ACC) and European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS) (ESC/EAS), and this part will not involve patient contact. Investigators will compare the P-CARDIAC risk score and the clinician's rating of a patient's recurrent CVD risk on a 10% random subgroup of patients from part one in a "silent deployment" approach, ie, an individual patient's P-CARDIAC risk score will not be communicated to cardiologists. Cardiologists will be invited to rate if they think the patient is at high or low risk according to existing risk scores and the proposed treatment management and target based on treatment guidelines based on their experience. Each patient profile will be reviewed by at least 2 cardiologists and discussed to reach a consensus. Investigators will then evaluate the sensitivity of P-CARDIAC risk score with clinician's judgment. Prior to the commencement of Part two, investigators will collect insights from cardiologists regarding the interpretability of performance metrics and acceptable threshold of model performance for clinical practice. In addition, through this exercise, the research team will assist cardiologists to draft a guideline for follow up for patients at different risk level.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 - 80 years old who visit the medical or cardiology SOPC clinics at the Queen Mary Hospital (QMH), Pok Oi Hospital (POH), Kwong Wah Hospital (KWH), Princess Margaret Hospital (PMH), Queen Elizabeth Hospital (QEH), Tuen Mun Hospital (TMH) and experienced prior CVD event (such as peripheral artery diseases, coronary heart diseases, myocardial infarction, stroke, revascularization) before the scheduled SOPC clinic visit date are eligible to participate in this study. Participants will be also able to comprehend English or Traditional Chinese as well.

Exclusion Criteria:

* People with history of dementia, psychiatric diseases or physical impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with established CVD visiting Queen Mary Hospital (QMH), Pok Oi Hospital (POH), Kwong Wah Hospital (KWH), Princess Margaret Hospital (PMH), Queen Elizabeth Hospital (QEH), Tuen Mun Hospital (TMH) during the study period will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
The relationship between P-CARDIAC risk score and heart disease related symptoms | From the date when participants join the project until the CVD outcomes confirmed in clinical setting or the date of death from any cause or the date of study ends whichever comes first, assessed up to 2 years.
  We hypothesize that patients with a higher frequency or larger number of types of cardiac event symptoms are likely to have a higher P-CARDIAC risk score. The correlation between P-CARDIAC risk score and the increasing in number of types and in number of times a patient reported to have heart disease symptoms, e.g. chest pain, shortness of breath, fatigue, swelling in legs, ankles or feet will be examined.
P-CARDIAC risk thresholds determination | From the date when participants join the project until the date of death from any cause or the study ends whichever comes first, accessed up to 2 years.
  The study will involve Delphi technique to determine P-CARDIAC risk thresholds with reference to current clinical management guideline such as American Heart Association (AHA)/American College of Cardiology (ACC) Multisociety Guideline (AHA/ACC) and European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS) (ESC/EAS), and this part will not involve paricipants contact.

CONTACTS AND LOCATIONS:
Overall Officials: Sze Ling Celine Chui, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhiting G, Jiaying T, Haiying H, Yuping Z, Qunfei Y, Jingfen J. Cardiovascular disease risk prediction models in the Chinese population- a systematic review and meta-analysis. BMC Public Health. 2022 Aug 24;22(1):1608. doi: 10.1186/s12889-022-13995-z. PMID 35999550
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Damman P, van 't Hof AW, Ten Berg JM, Jukema JW, Appelman Y, Liem AH, de Winter RJ. 2015 ESC guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: comments from the Dutch ACS working group. Neth Heart J. 2017 Mar;25(3):181-185. doi: 10.1007/s12471-016-0939-y. PMID 27966184
- [Background] Writing Committee Members; Drozda JP Jr, Ferguson TB Jr, Jneid H, Krumholz HM, Nallamothu BK, Olin JW, Ting HH; ACC/AHATask Force On Performance Measures; Heidenreich PA, Albert NM, Chan PS, Curtis LH, Ferguson TB Jr, Fonarow GC, Ho PM, O'Brien S, Russo AM, Thomas RJ, Ting HH, Varosy PD. 2015 ACC/AHA Focused Update of Secondary Prevention Lipid Performance Measures: A Report of the American College of Cardiology/American Heart Association Task Force on Performance Measures. Circ Cardiovasc Qual Outcomes. 2016 Jan;9(1):68-95. doi: 10.1161/HCQ.0000000000000014. Epub 2015 Dec 14. No abstract available. PMID 26666514
- [Background] Barrett D, Heale R. What are Delphi studies? Evid Based Nurs. 2020 Jul;23(3):68-69. doi: 10.1136/ebnurs-2020-103303. Epub 2020 May 19. No abstract available. PMID 32430290

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT06262828/Prot_SAP_000.pdf